CLINICAL TRIAL: NCT00002895
Title: A Randomised Trial in Relapsed Ovarian Cancer: Early Treatment Based on CA 125 Levels Alone Vs. Delayed Treatment Based On Conventional Clinical Indicators
Brief Title: Early Chemotherapy Based on CA 125 Level Alone Compared With Delayed Chemotherapy in Treating Patients With Recurrent Ovarian Epithelial , Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065218; MRC-OV05; EORTC-55955; ISRCTN87786644
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2005-09

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; primary peritoneal cavity cancer; fallopian tube cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Drug Therapy

INTERVENTIONS:
Drug: chemotherapy

SUMMARY:
RATIONALE: It is not yet known if treatment for recurrent ovarian epithelial, fallopian tube, or primary peritoneal cancer is more effective if it is begun when blood levels of CA 125 become elevated rather than waiting for other indicators of disease recurrence.

PURPOSE: This randomized phase III trial is studying early chemotherapy based on blood levels of CA 125 alone to see how well it works compared to chemotherapy based on conventional clinical indicators in patients with recurrent ovarian epithelial, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the benefit of early chemotherapy based on CA 125 level only vs chemotherapy based on conventional clinical indicators in patients with relapsed ovarian epithelial, fallopian tube, or primary peritoneal cancer.
* Compare the overall survival of patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients whose CA 125 levels rise to more than two times the upper limit of normal are randomized to one of two treatment arms.

* Arm I: The clinician is informed of the initial rise in CA 125 level. A confirmatory test is performed immediately. Within 4 weeks of the initial CA 125 elevation, patients with a second confirmed elevation receive treatment for recurrent disease according to standard local practice. Patients with a normal CA 125 on the confirmatory test receive no treatment until clinically indicated.
* Arm II: The clinician is blinded to the CA 125 results. Patients undergo normal monitoring. When clinically indicated, patients commence treatment according to standard local practice.

Quality of life is assessed at baseline, at each follow-up visit, and, if treatment is instituted, before each chemotherapy course.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 1,400 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, fallopian tube, or primary peritoneal cancer

  * Achieved complete remission with normal CA 125 after first-line platinum-containing chemotherapy
* Prior participation in the following clinical trials is allowed:

  * MRC-ICON2 (carboplatin vs cyclophosphamide, doxorubicin, and cisplatin for advanced disease)
  * MRC-ICON3 (paclitaxel with carboplatin in first-line therapy for advanced disease)
  * MRC-ICON5 (carboplatin and paclitaxel vs triplet and sequential doublet combinations of chemotherapy)
* No prior participation in MRC-ICON1 (adjuvant chemotherapy for early-stage ovarian cancer)

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No prior or concurrent malignancy within the past 5 years that is likely to preclude study treatment or comparisons except for nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 1996-06; Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Benefit of early chemotherapy
Overall survival
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Gordon J.S. Rustin, MD — Mount Vernon Cancer Centre at Mount Vernon Hospital; M. E.L. van der Burg, MD, PhD — University Medical Center Rotterdam at Erasmus Medical Center
Locations (21):
- Kaiser Franz Josef Hospital, Vienna, Austria
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - Cazk Groeninghe - Campus Maria's Voorzienigheid, Kortrijk
- Centre Regional Francois Baclesse, Caen, France
- Ireland (2):
  - Coombe Women's Hospital, Dublin
  - St. James' Hospital, Dublin
- Spedali Civili di Brescia, Brescia, Italy
- Netherlands (7):
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - Leiden University Medical Center, Leiden
  - Nijmegen Cancer Center at Radboud University Medical Center, Nijmegen
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
  - Leyenburg Ziekenhuis, The Hague
  - University Medical Center Utrecht, Utrecht
  - Isala Klinieken - locatie Sophia, Zwolle
- Hospitais da Universidade de Coimbra (HUC), Coimbra, Portugal
- Groote Schuur Hospital, Cape Town, South Africa
- Spain (3):
  - Institut d'Oncologia Corachan, Barcelona
  - Hospital Universitario San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England, United Kingdom

REFERENCES:
- [Background] Markman M, Petersen J, Belland A, Burg K. CA-125 monitoring in ovarian cancer: patient survey responses to the results of the MRC/EORTC CA-125 Surveillance Trial. Oncology. 2010;78(1):1-2. doi: 10.1159/000292352. Epub 2010 Mar 6. No abstract available. PMID 20215782
- [Result] Rustin GJ, van der Burg ME, Griffin CL, Guthrie D, Lamont A, Jayson GC, Kristensen G, Mediola C, Coens C, Qian W, Parmar MK, Swart AM; MRC OV05; EORTC 55955 investigators. Early versus delayed treatment of relapsed ovarian cancer (MRC OV05/EORTC 55955): a randomised trial. Lancet. 2010 Oct 2;376(9747):1155-63. doi: 10.1016/S0140-6736(10)61268-8. PMID 20888993
- [Result] Rustin GJ, van der Burg ME: A randomized trial in ovarian cancer (OC) of early treatment of relapse based on CA125 level alone versus delayed treatment based on conventional clinical indicators (MRC OV05/EORTC 55955 trials). [Abstract] J Clin Oncol 27 (Suppl 18): A-1, 2009.